CLINICAL TRIAL: NCT04628884
Title: Comparison of Two Strategies for Protamine Dosing After Anticoagulation in Cardiovascular Surgery Regarding Postoperative Bleeding: Total Heparin Administered Versus Residual Heparin Determined by a Pharmacokinetic Model
Brief Title: Strategies for Protamine Dosing After Anticoagulation in Cardiovascular Surgery
Acronym: SEPARATION
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundación Clínica Shaio (Other)
Collaborators: Universidad El Bosque, Bogotá (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DIB-20-34
Record Dates: First submitted 2020-11-09; First posted 2020-11-16 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Anticoagulant Antagonist Toxicity
Keywords: heparin; protamine; dose; extracorporeal circulation; cardiopulmonary bypass

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Protamine dosing according the total heparin administrated (Active Comparator): The protamine dose will be calculated according to the total heparin administered including the heparin dose add during the pump purge, 1 mg of protamine for each 100 IU of heparin
  Interventions: Drug: Conventional dose
- Protamine dosing according the residual heparin determined by a pharmacokinetic model (Experimental): The protamine dose will be calculated according to the residual heparin estimated before the separation of the cardiopulmonary bypass using a pharmacokinetic model, 1 mg of protamine for each 100 IU of residual heparin
  Interventions: Drug: Dosing according residual heparin

INTERVENTIONS:
Drug: Conventional dose — Conventional dose used to calculated the protamine dose
  Arms: Protamine dosing according the total heparin administrated
Drug: Dosing according residual heparin — In this group the heparin doses will be simulated using a pharmacokinetic model to estimated the residual heparin amount at the end of the surgery, the protamine dose will be calculated using the residual heparin
  Arms: Protamine dosing according the residual heparin determined by a pharmacokinetic model

SUMMARY:
In cardiovascular surgery, patients are anticoagulated with heparin during cardiopulmonary bypass, subsequently, anticoagulation is reversed with protamine to reduce bleeding due to residual heparin-induced coagulopathy, which can last more than four hours. Protamine reverses the effect of heparin by binding to each heparin molecule, therefore an amount of protamine equivalent to residual heparin is required at the time that anticoagulation is desired to be reversed, but generally, the dose of protamine is calculated from the total dose of heparin, ignoring that heparin is metabolized and cleared during of the extracorporeal circulation, this excess of protamine produces anticoagulant effects that increase postoperative bleeding. Residual heparin can be estimated from heparin pharmacokinetic models and therefore, from these models, a dose closer to the amount necessary to reverse the effect of heparin can be estimated, avoiding protamine excess. In this study, a protamine dosage strategy based on residual heparin determined by a pharmacokinetic model of heparin versus total administered heparin will be compared regarding bleeding and use of blood components in the postoperative period.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age who undergo scheduled cardiovascular surgery or scheduled urgency at the Shaio clinical foundation in the city of Bogotá, who require extracorporeal circulation.
* ASA classification, between 1 - 4
* Informed consent read and signed by the patient
* No history of known blood dyscrasia, with INR values <1.5
* Platelet count greater than 100,000
* No history of heparin-induced thrombocytopenia
* No history of adverse reaction to protamine
* No use of dual anti-aggregation therapy acetylsalicylic acid (ASA) + ADP receptor inhibitors (Clopidogrel) at the time of surgery
* Suspension of ADP receptor inhibitor drugs (Clopidogrel) according to institutional protocol.
* No use of bridging therapy with tirofiban
* Patient with chronic use of oral anticoagulants (warfarin, dabigatran), complete the suspension time according to the institutional protocol,
* No requirement for renal replacement therapy in the last month
* Patient with BMI between 18 - 41 kg / cm2
* Not pregnant

Exclusion Criteria:

* Emergency surgery
* Anticoagulated patient at the time of the intervention
* Procedure not performed under extracorporeal circulation.
* Procedure requiring circulatory arrest and / or profound hypothermia
* Intraoperative death before protamine administration
* Inability to complete data collection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2020-11-15 (Actual); Primary Completion 2021-11-20 (Estimated); Study Completion 2021-11-22 (Estimated)

PRIMARY OUTCOMES:
postoperative mediastinal bleeding | first 24 hours after surgery
  total blood collected from the mediastinal chest tubes during the first 24 hours

SECONDARY OUTCOMES:
total blood products transfused | first 24 hours after surgery
  red blood cells, plasma, cryoprecipitate, platelets, fibrinogen, and prothrombin complexes

CONTACTS AND LOCATIONS:
Overall Officials: Mauricio Abello, Study Chair — Fundacion Abood Shaio; David Ramez, Principal Investigator — Universidad del bosque
Locations (1):
- Fundacion Abood Shaio, Bogotá, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Puis L, Milojevic M, Boer C, De Somer FMJJ, Gudbjartsson T, van den Goor J, Jones TJ, Lomivorotov V, Merkle F, Ranucci M, Kunst G, Wahba A; EACTS/EACTA/EBCP Committee Reviewers. 2019 EACTS/EACTA/EBCP guidelines on cardiopulmonary bypass in adult cardiac surgery. Interact Cardiovasc Thorac Surg. 2020 Feb 1;30(2):161-202. doi: 10.1093/icvts/ivz251. No abstract available. PMID 31576402
- [Background] Delavenne X, Ollier E, Chollet S, Sandri F, Lanoiselee J, Hodin S, Montmartin A, Fuzellier JF, Mismetti P, Gergele L. Pharmacokinetic/pharmacodynamic model for unfractionated heparin dosing during cardiopulmonary bypass. Br J Anaesth. 2017 May 1;118(5):705-712. doi: 10.1093/bja/aex044. PMID 28510738
- [Background] Meesters MI, Veerhoek D, de Jong JR, Boer C. A Pharmacokinetic Model for Protamine Dosing After Cardiopulmonary Bypass. J Cardiothorac Vasc Anesth. 2016 Oct;30(5):1190-5. doi: 10.1053/j.jvca.2016.04.021. Epub 2016 Apr 28. PMID 27493093